CLINICAL TRIAL: NCT02448186
Title: Intervention Development for Social Stress, Mental Health, and HIV Risk Among MSM
Brief Title: Intervention Development for Social Stress, Mental Health, and HIV Risk MSM
Acronym: ESTEEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Hunter College of City University of New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1306012230
Record Dates: First submitted 2015-04-15; First posted 2015-05-19 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: HIV Infections; Depression; Anxiety
MeSH Terms: conditions — HIV Infections; Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ESTEEM (Experimental): cognitive behavioral treatment adapted to improve depression, anxiety, and co-occurring health risks (i.e., alcohol use, sexual compulsivity, condomless sex) among young adult gay and bisexual men by reducing minority stress processes that underlie sexual orientation-related mental health disparities
  Interventions: Behavioral: ESTEEM
- Waitlist (No Intervention): 3-month waitlist control

INTERVENTIONS:
Behavioral: ESTEEM — 10-session cognitive behavioral treatment
  Arms: ESTEEM

SUMMARY:
The proposed study will adapt a cognitive behavioral intervention to support high-risk MSM's adaptive coping with minority stress, alleviate associated depression and anxiety, and reduce HIV risk behavior. The adapted intervention is expected to increase awareness of the unhealthy impact of minority stress; facilitate objective self-schemas in the face of minority stress; and strengthen one's skills and self-efficacy for managing minority stress and associated anxiety and depression to reduce risk for acquiring HIV.

DETAILED DESCRIPTION:
Gay, bisexual, and other men who have sex with men (MSM) are the population most severely affected by HIV in the U.S. and one of the only risk groups in the U.S. for which new infections continue to rise. MSM also experience a vastly disproportionate risk of mental health disorders, especially depression and anxiety. Numerous studies have shown that this mental health disparity arises from the early and ongoing stressors, known as minority stress, that MSM experience related to their sexual orientation. Despite the fact that minority stress is strongly related to anxiety and depression, and that minority stress and related mental health problems synergistically propel HIV risk behaviors, no existing HIV prevention intervention targets minority stress in order to reduce MSM's HIV risk behavior. This project aims to develop a theoretically-driven intervention that reduces the health-depleting effects of minority stress through targeting the basic psychosocial mechanisms linking minority stress to HIV risk behavior. These mechanisms include maladaptive emotion regulation, negative thinking styles, low self-efficacy, avoidance, and impulsivity, which are the very targets of an existing cognitive-behavioral, manualized intervention--the Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders (UPTTED). The UPTTED changes these mechanisms using motivational interviewing, interoceptive and situational exposure, cognitive restructuring, mindfulness, and self-monitoring exercises, all grounded in cognitive-behavioral principles and developmental and affective neuroscience models of stress. The proposed study will adapt the UPTTED to support high-risk MSM's adaptive coping with minority stress, alleviate associated depression and anxiety, and reduce HIV risk behavior. The adapted UPTTED is expected to increase awareness of the unhealthy impact of minority stress; facilitate objective self-schemas in the face of minority stress; and strengthen one's skills and self-efficacy for managing minority stress and associated anxiety and depression to reduce risk for acquiring HIV. MSM who have experienced minority stress, mental health problems, and HIV risk behavior in the previous 3 months (n = 30) and community health experts (n = 30) will provide suggestions for adaptations to the existing intervention manual, including culturally relevant vignettes, examples, and exercises for adaptively responding to minority stress and managing HIV risk. The feasibility, acceptability, and preliminary efficacy of the adapted intervention will then be tested in a randomized waitlist controlled trial with MSM (n = 60) who report recent experiences with minority stress, depression and anxiety, and HIV risk behavior. The primary outcome will be HIV risk behavior. Secondary outcomes will be reductions in mediators including depression, anxiety, and the mechanisms of the conceptual model. This project innovatively seeks to test the preliminary efficacy of the first theoretically-driven intervention targeting the mental and sexual health consequences of minority stress and does so by targeting the underlying mechanisms that powerfully drive these simultaneous health threats.

ELIGIBILITY:
Inclusion Criteria:

1. Subjective stress related to sexual identity over the previous three months;
2. Symptoms of depression or anxiety within the past three months;
3. HIV sexual risk behavior (one or more acts of condomless insertive or receptive anal sex with a male partner of unknown or discordant serostatus) within the past three months;
4. Biological male gender;
5. At least 18 years of age;
6. Not known to have HIV;
7. Residential stability and availability for six months;
8. Ability to communicate in English; and
9. Provision of informed consent.

Exclusion Criteria:

1. active, unmedicated symptoms of bipolar I or bipolar II disorder or any Diagnostic and Statistical Manual-IV psychotic disorder in the past 12 months;
2. Current suicidal or homicidal ideation;
3. Evidence of gross cognitive impairment;
4. Current enrollment in an HIV-related intervention or research study; and
5. Knowledge of being infected with HIV.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2012-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
reductions in the number of condomless anal sex acts in the past 90 days with HIV-positive or HIV-status-unknown male partners | 3 months

SECONDARY OUTCOMES:
reduction in depression severity as measured with the Center for Epidemiological Studies Depression Scale | 3 months
reduction in anxiety severity as measured with the Overall Anxiety Severity & Impairment Scale | 3 months
reduction in minority stressors as measured with the Sexual Orientation Concealment Scale | 3 months
reductions in psychological risk factors measured with the Ruminative Responses Scale | 3 months
reductions in number of days in which heavy alcohol and potentially harmful recreational substances were use | 3 months
among individuals with body image disturbance, improvements in body attitudes as measured with the Male Body Attitude Scale | 3 months
among individuals with sexual compulsivity, reduction in sexual compulsivity severity as measured with the Sexual Compulsivity Scale | 3 months
reduction in alcohol use problems as assessed with the Alcohol Use Disorders Identification Test | 3 months
in participants with generalized anxiety disorder, reduction in Penn State Worry Questionnaire | 3 months
reduction in depression severity as measured with the Overall Depression Severity & Impairment Scale | 3 months
reduction in anxiety severity as measured with the State Trait Anxiety Inventory (State subscale) | 3 months
reduction in minority stressors as measured with the Internalized Homophobia Scale | 3 months
reduction in minority stressors as measured with the Rejection Sensitivity Scale | 3 months
reductions in psychological risk factors measured with the Rathus Assertiveness Schedule | 3 months
reductions in psychological risk factors measured with the Difficulties of Emotion Regulation Scale | 3 months
reductions in psychological risk factors measured with the Multidimensional Scale of Perceived Social Support | 3 months
in participants with obsessive-compulsive disorder, reductions in the Yale-Brown OC Scale | 3 months
in participants with panic disorder, reduction in the Panic Disorder Severity Scale | 3 months

REFERENCES:
- [Background] Pachankis JE. Uncovering Clinical Principles and Techniques to Address Minority Stress, Mental Health, and Related Health Risks Among Gay and Bisexual Men. Clin Psychol (New York). 2014 Dec;21(4):313-330. doi: 10.1111/cpsp.12078. PMID 25554721